CLINICAL TRIAL: NCT01378156
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of pGA2/JS7 DNA and MVA/HIV62B in HIV-infected Adults With Suppressed Viremia Who Started ART Within 18 Months of a Negative HIV Antibody Test
Brief Title: A Safety and Immunogenicity Study of a Plasmid DNA Prime and MVA Boost Vaccine in HIV-1 Infected Adults on ART
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GeoVax, Inc. (Industry)
Collaborators: AIDS Research Consortium of Atlanta (Other); University of Alabama at Birmingham (Other); AIDS Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GV-TH-01
Record Dates: First submitted 2010-07-30; First posted 2011-06-22 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: HIV-1 Infection
Keywords: Therapy for HIV Infection; Suppressive ART with no failures; Treatment interruption

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- JS7 plasmid DNA and MVA62B vaccines (Experimental): All subjects receive JS7 plasmid DNA (at 1 and 9 weeks) and MVA62B vaccines (17 and 25 weeks), followed (in 2 months after last vaccination) by a 12-week treatment interruption phase. Subjects reinstitute therapy after the treatment interruption and are followed for 6 months.
  Interventions: Biological: JS7 plasmid DNA and MVA62B vaccine

INTERVENTIONS:
Biological: JS7 plasmid DNA and MVA62B vaccine — JS7 plasmid DNA (3 mg at weeks 1 and 9) and MVA62B vaccine (10(8) TCID(50) at weeks 17 and 25)
  Other Names: pGA2/JS7 and MVA/HIV62B vaccine

SUMMARY:
GV-TH-01 is an open label Phase 1 study of 9 HIV-1 infected adults with suppressed viremia who started anti-retroviral therapy (ART) within 18 months of a negative HIV antibody test. This study has 3 phases. The first phase is the vaccination phase, where patients are vaccinated with pGA2/JS7 (JS7)DNA and MVA62B vaccines on a prime/boost regimen. The second phase of the study is a treatment interruption phase, whereby ART is interrupted for a 12 week period approximately 8 weeks following the last vaccination. The third phase occurs after the 12 week treatment interruption phase and is called the treatment reinstitution phase, because subjects reinstitute ART and are followed for an additional 24 weeks. The primary objective is to evaluate the safety of the vaccines during the three phases of the study. A secondary objective is to evaluate the immunogenicity of the vaccines during the vaccination phase of the study.

DETAILED DESCRIPTION:
GV-TH-01 is an open label Phase 1 study of 9 HIV-1 infected adults with suppressed viremia who started anti-retroviral therapy (ART) within 18 months of a negative HIV antibody test. This study has 3 phases. The first phase is the vaccination phase, where patients are vaccinated with pGA2/JS7 (JS7)DNA and MVA62B vaccines on a prime/boost regimen at weeks 1 and 9 (JS7 DNA vaccine) and weeks 17 and 25 (MVA62B). Both vaccines express Gag, Pol, and Env. The second phase of the study is a treatment interruption phase, whereby ART is interrupted for a 12 week period approximately 8 weeks following the last vaccination. The third phase occurs after the 12 week treatment interruption phase and is called the treatment reinstitution phase, because subjects reinstitute ART and are followed for an additional 24 weeks. The primary objective is to evaluate the safety of the vaccines during the three phases of the study. A secondary objective is to evaluate the immunogenicity of the vaccines during the vaccination phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 yrs.
* ART started within 18 mo. of last documented negative HIV Ab test, or within 13 mo. of last negative detuned HIV-1 Ab assay, or within 18 mo. of evolution of Western blot from indeterminate to positive in the presence of a positive Ab test
* No changes to ART treatment within 4 wks. of study entry
* Documentation of level of plasma HIV-1 RNA and CD4+ counts prior to ART
* On stable suppressive ART [HIV-1 RNA < 50 copies/mL (PCR) or < 75 copies/mL (bDNA) for at least 6 mo. prior to starting vaccination]
* No history of virologic failure
* CD4+ > 500 cells/µL
* Nadir CD4+ > 350 cells/µL unless measured in the setting of acute infection
* Laboratory values:

  * Hemoglobin ≥ 10g/dL (male) or 9g/dL (women)
  * ANC > 1000 cells/µL
  * ALT, AST ≤ 2.5 ULN
  * Total bilirubin < 1.5 x ULN (≤ 5 x ULN on atazanavir)
  * Fasting glucose ≤ 125 mg/dL
  * Serum creatine < 1.5 x ULN
  * Creatinine clearance ≥ 60 mL/min (Cockcroft-Gault)
  * Serum creatine phosphokinase (CPK) ≤ 1.5 x ULN
  * UA negative for hemoglobin and glucose and no greater than 1+ protein
  * Any abnormalities must be assessed by the investigator as not clinically significant
* ECG without evidence of current or past MI, or ischemic heart disease
* Willing to provide signed informed consent
* Females: a negative serum or urine β-HCG pregnancy test at screening
* Female subjects of reproductive potential who engage in sexual activity that could lead to pregnancy must agree to avoid pregnancy and agree to consistently use contraception for at least 21 days prior to first vaccination until the last protocol visit.
* Male subjects participating in the study must agree to not attempt to impregnate a female, or participate in sperm donation programs
* Males engaging in sexual activity that could lead to pregnancy must use a condom from the date of receipt of the first study vaccine until the last protocol visit
* Agreement to use condoms for protection against HIV-1 transmission throughout the study
* Participants must be willing to comply with all study requirements and expected to be available for the duration of the study
* Participants must be willing to temporarily discontinue antiretroviral therapy for up to 12 wks. post-vaccinations

Exclusion Criteria:

* Known infection with HIV-1 subtype other than Clade B
* Chemotherapy for active malignancy in the past 12 mo.
* Prior vaccinations with any HIV-1 vaccine
* Prior vaccination against smallpox within the last 15 yrs.
* History of or known cardiac disease
* History of myositis
* Diagnosis of HIV-associated nephropathy
* Evidence of active HBV or HCV infection
* Framingham Global Risk Assessment Score consistent with high short-term (10 yr.) cardiac risk
* Receipt of immunomodulatory agents, systemic corticosteroids (including nonprescription street steroids), gamma globulin, or investigational agents (other than H1N1 influenza vaccine) within 6 mo. of screening
* Any immunization within 1 mo. of screening and within 2 wks. of any inoculation in this study
* Creatine supplements within 14 days of baseline and unwillingness to discontinue use throughout the trial
* Changes in ART regimen prior to entry due to virologic failure (not including toxicity)
* Pregnancy or breastfeeding
* Any clinically significant diseases (other than HIV-1 infection) or clinically significant findings during the screening medical history or physical examination that, in the investigator's opinion, would compromise participant safety
* Active alcohol or substance abuses
* Allergy to chicken egg derived products
* Contraindication to intramuscular injection
* Unwilling to forego vigorous exercise 3 days prior to each vaccination

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2010-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Safety in all phases of study. | Throughout study - up to 77 weeks
  Frequency and severity of adverse events, laboratory abnormalities, and local and systemic reactogenicity signs and symptoms following vaccinations. Vaccination(virologic failure): HIV-1 RNA >200 copies/mL and CD4+ <350 cells/uL; genotypic resistance patterns of re-emergent virus. Treatment interruption:number(#)and percentage(%): 1)meet HIV-1 RNA and CD4+ criteria to re-institute anti-retroviral therapy before 12 wks; 2)genotypic resistance in re-emergent virus. Treatment reinstitution:# and %: 1)meet criteria for virologic failure; 2)genotypic resistance in patients with virologic failure.

SECONDARY OUTCOMES:
Immunogenicity | Throughout vaccination and treatment interruption phases
  Magnitude of interferon (ifn) gamma &/or interleukin-2 (IL-2) producing CD4+ and CD8+ T cells at 1 week (wk) post 2nd MVA (modified vaccinia ankara) vaccination (vacc); titer & avidity index of binding aby for Env at 2 wks post 2nd MVA vacc. Magnitude of ifn-gamma &/or IL-2 producing CD4+ & CD8+ cells, # and id of Gag-specific CD8+ responses & titers of binding aby for Env at 2 wks post detection of re-emergent virus. Log change in HIV-1 RNA from before antiretroviral therapy to end of treatment interruption; time to HIV-1 rebound to >200 copies/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Harriet L Robinson, PhD, Study Chair — GeoVax, Inc.
Locations (3):
- United States (3):
  - The University of Alabama at Birmingham Alabama Vaccine Research Clinic, Birmingham, Alabama
  - AIDS Research Alliance, Los Angeles, California
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia

REFERENCES:
- [Result] Thompson M, Heath SL, Sweeton B, Williams K, Cunningham P, Keele BF, Sen S, Palmer BE, Chomont N, Xu Y, Basu R, Hellerstein MS, Kwa S, Robinson HL. DNA/MVA Vaccination of HIV-1 Infected Participants with Viral Suppression on Antiretroviral Therapy, followed by Treatment Interruption: Elicitation of Immune Responses without Control of Re-Emergent Virus. PLoS One. 2016 Oct 6;11(10):e0163164. doi: 10.1371/journal.pone.0163164. eCollection 2016. PMID 27711228